CLINICAL TRIAL: NCT02299154
Title: Study of Memory Problems Perceptions With the French Adaptation of the Illness Perception Questionnaire Memory, Among Patients Who Come for the First Time at a Memory Center Until Diagnosis Disclosure Post-visit
Brief Title: Memory Problems Perceptions Among Patients and Accompaniers During Diagnosis Process :
Acronym: REMAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: France Alzheimer (Other); Laboratoire APEMAC :Maladies chroniques, santé perçue, processus d adaptation, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00156-41
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Memory Disorders; Alzheimer Disease
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with memory disorders (Experimental): psychological questionnaires
  Interventions: Behavioral: Psychological questionnaires
- Accompanier (Experimental): psychological questionnaires
  Interventions: Behavioral: Psychological questionnaires

INTERVENTIONS:
Behavioral: Psychological questionnaires — Psychological questionnaires about memory problems perceptions, anxiety, depression, quality of life and coping

SUMMARY:
This study aims to prospectively examine the memory problem perceptions of patients with memory complaints [MCs] and their accompaniers during the diagnostic process.

DETAILED DESCRIPTION:
Through the french adaptation of the "illness perception questionnaire memory", this study aims to prospectively examine the memory problem perceptions of patients with memory complaints [MCs] and their accompaniers during the diagnostic process. The investigators plan to recruit 125 patients with MCs who come for the first time at the Research and Resources Memory Center in Nancy, France. Participants have to express MCs and must be free of dementia diagnosis at the first visit. Participants also need to be accompanied by an accompanier and both have to be fluent in French. This study has been approved by our local Ethics Committee (Committee for the Protection of Persons) and the French Health Security Agency. After giving their informed consent, patients and accompaniers are followed up throughout the diagnostic process with three visits : at their first visit, at one month after the first visit, and at six months after the diagnosis disclosure.

ELIGIBILITY:
Inclusion Criteria:

For patients with memory complaints:

* Age over 18 years
* Have a memory complaints with a QPC score greater than or equal to 3
* Be accompanied by a next of kin
* Folstein MMSE greater than or equal to 15/30
* Have given their written consent after receiving clear and intelligible oral and written information
* Social security coverage

For Accompaniers :

* Age over 18 years
* Consent to participate at the study with the patient
* Have given their written consent after receiving clear and intelligible oral and written information
* Social security coverage
* Be in contact with the patient at least 8 hours per week. It could be physical contact or telephone contact.

Exclusion Criteria:

For patients with memory complaints:

* Sensory deficit interfering with the completion of the questionnaires
* Level of French insufficient to complete the questionnaires
* Legally protected person
* Diagnosis of neurocognitive disorders already established
* Treatment for Alzheimer Disease
* Refusal or inability to obtain written informed consent form from the patient
* Included in another experimental study at inclusion visit

For Accompaniers:

* Sensory deficit interfering with the completion of the questionnaires
* Level of French insufficient to complete the questionnaires
* Refusal or inability to obtain written informed consent form from the accompanier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Memory problems perceptions of patients and next of kin during diagnosis process | Baseline and 6 months after diagnosis disclosure
  How patients and accompaniers perceive memory problems at the first visit in a Memory Center to 6 months after the diagnosis disclosure, with the Illness Perception Questionnaire Memory

SECONDARY OUTCOMES:
Psychometric properties of the french adaptation of the Ilness Perceptions Questionnaire - Memory (IPQ-M, Hurt et al. 2010) | Baseline, 1 month later and 6 months after diagnosis disclosure
  Psychometric properties of IPQ-M by a traditional approach and by comparison to another french memory complaint questionnaire
Impact of the memory problems perceptions on mood and well-being | Baseline and 6 months after diagnosis disclosure
  Correlation between memory problems perceptions at the IPQ-M, levels of anxiety (STAI-Y), depression (MADRS), quality of life (WHOQOL-BREF) and coping strategies.
Differences of memory problems perceptions and coping according to level of cognitive disorder at the Mini-Mental State Examination (MMSE) | Baseline and 6 months after diagnosis disclosure

CONTACTS AND LOCATIONS:
Overall Officials: Christine Perret-Guillaume, PhD, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- University Hospital of Nancy ,CHU Brabois, France, Vandœuvre-lès-Nancy, France